CLINICAL TRIAL: NCT03193073
Title: Impact of Anemia Correction and Fibroblast Growth Factor 23 Levels in Left Ventricular Hypertrophy, and Early Endothelial Dysfunction in Chronic Kidney Disease, and Renal Transplant Patient
Brief Title: Anemia Correction and Fibroblast Growth Factor 23 Levels in Chronic Kidney Disease , and Renal Transplant Patient
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: problem in funding which will be solved by the end of August
Sponsor: Omnia Mohammed Hashem (Other)
Responsible Party: Sponsor-Investigator, Omnia Mohammed Hashem, Assistant lecturer at Assiuy university- faculty of medicine-internal medicine department, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17200031
Record Dates: First submitted 2017-05-26; First posted 2017-06-20 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Anemia of Chronic Kidney Disease; Endothelial Dysfunction; Left Ventricular Hypertrophy; Fibroblast Growth Factor 23
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Intervention Model Description: two groups of patients (group A: CKD and group B newly transplanted patients) are assigned for detailed echocardiography , serum FGF-23, flow mediated dilatation of the forearm before anaemia correction in group A and renal transplant in group B .
  Also assesment of FGF-23 in different stages of group A, assessment of FGF-23 before and after renal transplant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD patients with different stages (Active Comparator): 1. Full clinical history and through clinical examination.
  2. Full blood count at time of diagnosis and 3 months after initiation of treatment with iron and erythropoietin Stimulating agents.
  3. Iron study at time of diagnosis and 3 months after treatment .
  4. Serum calcium , phosphorus, intact Parathrmone hormone. 5-24- urinary proteins or Albumin Creatinine ratio every month (for 3 months )then every 3 months (1 st year), then annually.
  6- Lipid profile . 7-Estimated glomerular filtration rate by MDRD equation .
  Interventions: Diagnostic Test: detailed echocardiography; Diagnostic Test: serum fibroblast growth factor-23; Diagnostic Test: flow mediated dilatation of forearm
- Newly renal transplanted patients . (Active Comparator): 1. Full clinical history and through clinical examination.
  2. Pre transplant Serum calcium , phosphorus , I Parathrmone hormone , serial measures every / 3 months for 2 years.
  3. Pre-transplant full blood count serial measures every / 3 months for 2 years.
  4. Pre transplant serum Iron study and annually for 2 years.
  5. 24- urinary proteins or albumin-creatinine ratio every month (for 3 months )then every 3 months (1 st year), then annually.
  6. Post-transplant serum FGF-23 (as independent risk factor) at 6months.
  7. Different immunosuppressive protocols.
  8. Pre-transplant panel reactive antibody,donor-specific antibody
  Interventions: Diagnostic Test: detailed echocardiography; Diagnostic Test: serum fibroblast growth factor-23; Diagnostic Test: flow mediated dilatation of forearm

INTERVENTIONS:
Diagnostic Test: detailed echocardiography — Detailed Echocardiography including ejection fraction, interventricular septum thickness, posterior wall thickness, left ventricular end -diastolic and end- systolic diameter and left ventricular mass index will be correlated with body surface area for both groups serum FGF-23
Diagnostic Test: serum fibroblast growth factor-23 — serum levels of FGF-23
Diagnostic Test: flow mediated dilatation of forearm — superficial sonar assess the diameter of brachial vessel on exposure to stress

SUMMARY:
The fibroblast growth factor-23-bone-kidney axis is part of newly discovered biological systems linking bone to other organ functions through a complex endocrine network that is integrated with the parathormone/vitamin D axis and which plays an equally important role in health and disease . Most of the known physiological function of fibroblast growth factor 23 to regulate mineral metabolism can be accounted for by actions of this hormone on the kidney.In a recent experimental study, fibroblast growth factor-23 was shown to cause pathological hypertrophy in rat cardiomyocytes by "calcineurin-nuclear factor of activated T cells" and treatment with fibroblast growth factor -blockers reduced left ventricular hypertrophy in experimental models of chronic renal failure.The current hypothesis is that, in healthy individuals, iron deficiency stimulates increased production of fibroblast growth factor23. At the same time, iron is thought to be the cofactor of enzymes taking part in the degradation of intact fibroblast growth factor-23 and thought to have a role in the excretion of degraded FGF-23 parts .Studies speculated that Angiotensin Converting Enzyme inhibitors may exert their anti-proteinuria effects at least in part by reducing serum fibroblast growth factor-23 levels although it is difficult from the results of this study to understand which comes first and brings about the other; decrease in proteinuria or fibroblast growth factor-23. Available evidence points to the deleterious effects of increased fibroblast growth factor-23 level in proteinuria, but the precise molecular mechanism still remains to be explored. An intricate and close association exists among parathormone, phosphorus, active vitamin D with FGF23, but the independent role of the latter on proteinuria is the least explored. Elaborately conducted studies that control effects of confounding factors adequately are needed to demonstrate the independent pathogenic role of FGF23.

DETAILED DESCRIPTION:
1. To study the effect of anemia correction and left ventricular hypertrophy in Chronic Kidney Disease patients and renal transplant patients .
2. To study the relation of fibroblast growth factor and Left ventricular hypertrophy in Chronic kidney disease and renal transplant patients.
3. To study the relation between fibroblast growth factor 23 and early endothelial dysfunction in both Chronic kidney disease and renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

All patients:

1. Above 18 years old
2. Diagnosed as CKD, and renal transplanted patients at Assiut University Hospital in the period 2017-2020 .

Exclusion Criteria:

1. Severely hypocalcaemic patients < 7mg/dl.
2. Severely hyperphosphatemic patients >7 mg/dl .
3. Uncontrolled hypertensive patients ( more than 3 antihypertensive drugs).
4. Uncontrolled diabetic patients HBA1C >8 .
5. Blood transfusion dependent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
if change of in Hemoglobin level and correction of anemia associated with change in the left ventricular outcomes | measures at time of diagnosis then after 3 months
  measure the left ventricular mass index (gm/m2)
the relationship between the FGF-23 and degree of left ventricular dysfunction | measure at time of diagnosis
  measure FGF-23 level in (pg/ml)
the relationship between FGF-23 level and early endothelial dysfunction | at time of diagnosis in chronic kidney disease / after 6 months in renal transplant
  change in arterial diameter in mm

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Ali Tohamy, professor, Study Director — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Grabner A, Amaral AP, Schramm K, Singh S, Sloan A, Yanucil C, Li J, Shehadeh LA, Hare JM, David V, Martin A, Fornoni A, Di Marco GS, Kentrup D, Reuter S, Mayer AB, Pavenstadt H, Stypmann J, Kuhn C, Hille S, Frey N, Leifheit-Nestler M, Richter B, Haffner D, Abraham R, Bange J, Sperl B, Ullrich A, Brand M, Wolf M, Faul C. Activation of Cardiac Fibroblast Growth Factor Receptor 4 Causes Left Ventricular Hypertrophy. Cell Metab. 2015 Dec 1;22(6):1020-32. doi: 10.1016/j.cmet.2015.09.002. Epub 2015 Oct 1. PMID 26437603
- [Result] Torun D, Yildiz I, Micozkadioglu H, Nursal GN, Yigit F, Ozelsancak R. The effects of cinacalcet treatment on bone mineral metabolism, anemia parameters, left ventricular mass index and parathyroid gland volume in hemodialysis patients with severe secondary hyperparathyroidism. Saudi J Kidney Dis Transpl. 2016 Jan;27(1):15-22. doi: 10.4103/1319-2442.174053. PMID 26787561
- [Result] Wolf M, Koch TA, Bregman DB. Effects of iron deficiency anemia and its treatment on fibroblast growth factor 23 and phosphate homeostasis in women. J Bone Miner Res. 2013 Aug;28(8):1793-803. doi: 10.1002/jbmr.1923. PMID 23505057
- [Result] Eser B, Yayar O, Buyukbakkal M, Erdogan B, Ercan Z, Merhametsiz O, Haspulat A, Oguz EG, Dogan I, Canbakan B, Ayli MD. Fibroblast growth factor is associated to left ventricular mass index, anemia and low values of transferrin saturation. Nefrologia. 2015;35(5):465-72. doi: 10.1016/j.nefro.2015.06.025. Epub 2015 Sep 26. English, Spanish. PMID 26394828
- [Result] Io H, Aizawa M, Funabiki K, Horikoshi S, Tomino Y. Impact of anaemia treatment for left ventricular remodelling prior to initiation of dialysis in chronic kidney disease patients: Efficacy and stability of long acting erythropoietin stimulating agents. Nephrology (Carlton). 2015 Dec;20 Suppl 4:7-13. doi: 10.1111/nep.12640. PMID 26439537